CLINICAL TRIAL: NCT04713345
Title: VERARE_2 Efficacy of the Observation of Virtual Motor Actions for the Improvement of Gait in Patients With ICU Weakness
Brief Title: VERARE_2 Efficacy of the Observation of Virtual Motor Actions for the Improvement of Gait in Patients With ICU-weakness
Acronym: VERARE_2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Collaborators: Equipe Hybrid, INRIA - Campus Universitaire de Beaulieu - F-35042 Rennes Cedex - France (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 35RC20_3078_VERARE_2; 2020-A03462-37 (Other: ID RCB)
Record Dates: First submitted 2020-12-14; First posted 2021-01-19 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: ICU-weakness
Keywords: resuscitation; ICU-weakness; virtual reality; avatar; rehabilitation

STUDY DESIGN:
Intervention Model Description: Pilot, single-center, prospective, randomized, open-label, superiority study with 2 parallel groups (1: 1): experimental group (Virtual Reality) versus control group (Relaxation).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): If the patient is included in the Virtual Reality group, they will be asked to observe 1 time per day for 9 days for 5 minutes Virtual Motor Actions (avatar moving in a virtual environment) using a headset. Virtual Reality, followed by 5 minutes of relaxation performed using soothing music played through headphones.
  Interventions: Other: Virtual Reality Observations
- Control group (Sham Comparator): If the patient is included in the Relaxation group, they will be offered 10 minutes of relaxation performed using soothing music played through headphones once a day for 9 days.
  Interventions: Other: Relaxation

INTERVENTIONS:
Other: Virtual Reality Observations — If the patient is included in the Virtual Reality group, they will be asked to observe 1 time per day for 9 days for 5 minutes Virtual Motor Actions (avatar moving in a virtual environment) using a headset. Virtual Reality, followed by 5 minutes of relaxation performed using soothing music played through headphones.
  Arms: Experimental group
Other: Relaxation — If the patient is included in the Relaxation group, they will be offered 10 minutes of relaxation performed using soothing music played through headphones once a day for 9 days.
  Arms: Control group

SUMMARY:
After hospitalization in Intensive Care (Intensive Care Unit or Continuing Care Unit), approximately 50% of patients usually present with intensive ICU-weakness, i.e. damage to the nerves and muscles secondary to immobilization and to the treatments that must have been used. This condition will delay the resumption of walking in these patients, their discharge from hospital and impair their autonomy in the daily life.

The recent international literature is in favor of early rehabilitative management of these patients, which should ideally be started in the intensive care unit. However, this is not always possible, due to the possible lack of physiotherapists in the services on the one hand, due to the fatigue of the population concerned and the existence of unstable medical conditions which do not always allow the use of recommended rehabilitation techniques on the other hand.

Virtual Reality (VR) environments are widely used for the assessment and rehabilitation of patients with neurological pathology. VR allows the user to be active in simulated activities and offers many advantages for the rehabilitation of motor functions in patients with neurological diseases. VR tools used to create action observation, motor imagery and sensations or even the illusion of movement in particular, have already shown their effectiveness in recovering and improving walking in different populations, especially after a stroke, in patients with Parkinson's Disease or Multiple Sclerosis. The role of the embodiment in VR appears promising in immersing participants in a controlled environment and creating movement's illusions.

The Virtual Reality tool designed consists of virtual environments presented using a Virtual Reality headset where an avatar (double) of the hospitalized patient will be represented, who will perform a walking motor task (involving his lower limbs ) in several different virtual environments (sets). In the present study named VERARE_2, the patient will be asked to observe walking actions and imagine performing them as they will be performed by the avatar in the virtual environment.

This VERARE_2 protocol aims to assess the effectiveness of the Observation of Virtual Motor Actions on the speed of gait recovery in hospitalized patients with IUC-weakness and in the intensive care units and continuing care units of the Rennes University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized in one of the ICU or Continuing Care Units or at the CHU de Rennes for less than 3 months, and presenting lower limb muscle weakness with MRC motor testing on the main muscle segments giving a score of less than or equal to 48/60 (ICU Weakness diagnostic criterion) in the aftermath of severe sepsis.
* Person of full age;
* Affiliation to a social security scheme;
* Free, informed and signed written consent.

Exclusion Criteria:

* History of a central neurological event with clinical repercussions
* Gait disorders pre-existing to hospitalization in intensive care and limiting the walking perimeter (declaration by the patient) or requiring the use of technical assistance;
* Uncontrolled epilepsy (seizure less than 6 months old);
* Adults who are the subject of legal protection (safeguard of justice, curatorship, guardianship), persons deprived of their liberty;
* Non-French speaking person;
* Pregnant or breastfeeding woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2025-09-02 (Estimated)

PRIMARY OUTCOMES:
6-minute walking test | Day 9
  Number of meters taken during the 6-minute test the day after the last session

SECONDARY OUTCOMES:
10-meter walking test | Day1, day 9, month 1 and month 3
  Assessment of walking before the start of the first session, the day after the last session and 1 month after inclusion: 10-meter test (time in seconds)
6-minute walking test | Day1, day 9, month 1 and month 3
  Assessment of walking before the start of the first session, the day after the last session and 1 month after inclusion: 6-minute walk test (need for breaks, scale of Borg, existence of a desaturation)
Recovery time | Day 1, day 9, month 1 and month 3
  Assessment of walking before the start of the first session, the day after the last session and 1 month after inclusion: recovery time of walking over 10 meters without human or technical assistance
Berg Balance Scale | Day 1, day 9, month 1 and month 3
  Balance assessment before the start of the first session, the day after the last session and 1 month from inclusion: Berg Balance Scale Berg's Balance Rating Scale consists of 14 tests that assess static and dynamic balance.
  Static balance (standing without movement of the feet) is measured by the following tasks:
  Feet glued together Unipodal support Tandem (one foot in front of the other) Eyes closed Trunk rotation
  Dynamic balance is measured by the following tasks:
  360º swivel Pick up an object Get up and sit down Seated transfer from one chair to another
  All items except one are performed standing. They are rated on a 5-point ordinal scale (0-4) based on the ability to perform the movement or task independently, and criteria of time and distance. The total score varies between 0 and 56 points; a high score corresponds to a better balance [3, 4]. A score of 0 to 20 is associated with disturbed balance, 21 to 40 for acceptable balance and 41 to 56 for good balance.
Timed Up and Go test | Day 1, day 9, month 1 and month 3
  Balance assessment before the start of the first session, the day after the last session and 1 month from inclusion: Timed Up and Go test (time in seconds)
Test of the 10 chair lifts | Day 1, day 9, month 1 and month 3
  Balance assessment before the start of the first session, the day after the last session and 1 month from inclusion: test of the 10 chair lifts (duration in seconds, existence of a desaturation, Borg scale)
Strength | Day 1, day 9, month 1 and month 3
  Strength assessment before the start of the first session, the day after the last session and 1 month after inclusion: MRC (Medical research council) testing of the lower limbs
  0 No muscle contraction.
  1. Muscle contraction without movement.
  2. Movement in the plane of the bed.
  3. Movement against gravity.
  4. Movement against resistance.
  5. Normal muscle strength.
Force | Day 1, day 9, month 1 and month 3
  3 manual dynamometer force measurements per upper limb
Autonomy | Day 1, day 9, month 1 and month 3
  Assessment of autonomy before the start of the first session, the day after the last session and 1 month from inclusion using the FIM (Functional Independence Measure) FIM scores range from 1 to 7. The grading categories range from "total assistance with helper = 1" to "complete independence with no helper=7.
Confidence | Day 1, day 9, month 1 and month 3
  Assessment of confidence in the future using a questionnaire before the start of the first session, the day after the last session, 1 month after inclusion and 3 months after inclusion.
Recovery time | Month 1
  Assessment of the recovery time from a possible 10-meter walk without human or technical assistance in this population (in days between the day of hospitalization in intensive care and the day of recovery from a possible 10-meter walk without human assistance neither technique, a criterion which is noted in the patient's medical file by his physiotherapist in current clinical practice)
Acceptance | Day 9
  Acceptance questionnaire (established by the sponsor) : 54 items ranged from 1 to 7 (1 : not at all; 7 : completely) and 1 grade out of 10 and 1 to percentage
Tiredness | Days 1, 2, 3, 4, 5, 6, 7 and 8
  Assessment of tiredness using a Visual Analogue Scale (VAS) from 0 = no fatigue to 7 = intense fatigue, at the end of each session with the Virtual Reality tool
Rate of Adverse effects | Days 1, 2, 3, 4, 5, 6, 7 and 8
  Number of participants reporting any adverse effect during the intervention by open question at the end of each session with the Virtual Reality tool

CONTACTS AND LOCATIONS:
Locations (1):
- Rennes University Hospital, Rennes, Brittany Region, France